CLINICAL TRIAL: NCT00355251
Title: Study of the Influence of Atorvastatin in Plasma Viral Replication Given Prior to Antiretroviral Treatment Interruption in Patients With HIV-1 Infection and Viral Suppression.
Brief Title: Influence of Atorvastatin on Viral Replication During Antiretroviral Treatment Interruption
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: On the basis of published results of SMART study, it has been observed that the results are worse in patients who have interrupted their treatments.
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Fundació Lluita contra la Sida, Fundació Lluita contra la Sida
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRE-ATOR; 2005-005356-41
Record Dates: First submitted 2006-07-19; First posted 2006-07-21 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-02

CONDITIONS: HIV Infections
Keywords: Atorvastatin; Viral replication; HIV-1; plasma cholesterol; Cell membrane cholesterol
MeSH Terms: conditions — HIV Infections | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 4 semanas manteniendo el tratamiento antirretroviral e iniciar atorvastatina 40 mg/día. A la semana 4 interrupción HAART y aumentar a 80 mg/día de atorvastatina hasta la semana 32 de seguimiento
  Interventions: Drug: Atorvastatin 40 mg/Atorvastatin 80 mg
- B (No Intervention): 4 semanas manteniendo el tratamiento antirretroviral. A la semana 4 interrupción HAART hasta la semana 32 de seguimiento

INTERVENTIONS:
Drug: Atorvastatin 40 mg/Atorvastatin 80 mg — Atorvastatin 40 mg/80 mg
  Arms: A

SUMMARY:
To determine the influence of atorvastatin on plasma viral replication when the latter is given before and during highly active anti-retroviral therapy (HAART) in patients with HIV infection and viral suppression.

DETAILED DESCRIPTION:
Recently, the inhibitory effect of the statins on the replication of the human immunodeficiency virus Type 1 (HIV-1) through two independent mechanisms of action has been described: the blockade of Rho guanosine triphosphatase that intervenes in the entry and exit of the virus and the blockade of the interaction between LFA-1 (leukocyte function antigen 1) and its ICAM 1 ligand (intercellular adhesion molecule 1) that intervenes in the process through which the virus binds to the target cell.

These initial data have led to the study of the effect of atorvastatin on the plasma replication of HIV in HIV+ patients that interrupt antiretroviral therapy (Ator Study 3) developed in our unit. The data of this study indicate that baseline plasma cholesterol determines viral load rebound on interrupting antiretroviral treatment. However, the introduction of atorvastatin on the day of interruption provided no virological or immunological benefit in comparison with an interruption of antiretrovirals without statins. This may be due to the fact that the potent inhibitory effect of atorvastatin is unable to compensate their activating effect on the production of HIV also described in our study.

Overall, our results pose a possible usefulness of atorvastatin in the control of viral replication if given before the interruption of antiretroviral therapy due to:

* Their capacity to reduce serum cholesterol at the time of interruption and consequently the cholesterol of the cell membrane.
* Their potent capacity to purge the HIV reservoir

Therefore, in this study we aim to investigate the impact of atorvastatin on viral replication when it is given 8 weeks before the interruption of the antiretroviral treatment and determine whether this impact is due to the reduction in serum and/or membrane cholesterol, or whether, on the other hand, there is a contribution by atorvastatin's capacity to induce the expression of viral products.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years.
2. Patients with chronic infection by HIV-1 in stable highly active antiretroviral treatment (>= 6 months).
3. Undetectable plasma viral load (<50 copies/mL) in the last 3 determinations over the last 6 months.
4. CD4 > 500 cells/mm>=3 in the last two determinations.
5. Documented prior viral load at some time of >15,000 copies/mL.
6. Women may not be of fertile age (defined as at least one year from menopause or undergoing any surgical sterilisation technique), or must undertake to use a barrier contraceptive method during the study.
7. Signature of the informed consent

Exclusion Criteria:

1. CD4 nadir <= 200 cells/mm3.
2. Background of infections or other AIDS-defining pathology.
3. Intercurrent infections in the last 6 months.
4. Creatine kinase (CK) >= 500 U/L.
5. AST or ALT >= 3 times higher than the upper limit of normality.
6. Treatment with others statins, fibrates, macrolides or fluconazole in the last 3 months.
7. Pregnancy or breastfeeding
8. Patients participating in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-07; Primary Completion 2006-12 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is viral load (HIV RNA) in plasma. | at 12 and 24 weeks

SECONDARY OUTCOMES:
CD4 and CD8, absolute value, percentage and activation. | during the 32 weeks of follow-up
Total cholesterol, HDL and LDL in serum. | during the 32 weeks of follow-up
Cholesterol in cell membrane. | during the 32 weeks of follow-up
Symptoms reported by the patient following the interruption of the HAART therapy or signs detected by the clinician (classification according to the WHO), mainly those which may indicate acute antiretroviral symptoms. | during the 32 weeks of follow-up
Creatinine, urea, creatine kinase (CK), hepatic tests, (AST, ALT, GGT) | during the 32 weeks of follow-up
Proviral load. | during the 32 weeks of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventura Clotet, MD,PhD, Principal Investigator — LLuita contra la Sida Foundation-HIV Unit
Locations (1):
- Germans Trias i Pujol Hospital, Badalona, Barcelona, Spain